CLINICAL TRIAL: NCT01788371
Title: Nucleoside Analogue in Late Preganancy to Prevent Vertical Transmission of Hepatitis B Virus
Brief Title: Nucleoside Analogue Prevent Vertical Transmission of Hepatitis B Virus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hua Zhang (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor-Investigator, Hua Zhang, Professor, Beijing YouAn Hospital
Organization: Beijing YouAn Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2011.6
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Hepatitis B Infection; Chronic Infection; Viremia
MeSH Terms: conditions — Hepatitis B; Persistent Infection; Viremia | interventions — Telbivudine; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- No antiviral arm (No Intervention): provide standard of care to mothers and standard immunoprophylaxis to their infants
- Lamivudine (Experimental): lamivudine treatment from 28 weeks of pregancy to week 4 of postpartum for mothers and standrd immunoprophylaxis to their infants
  Interventions: Drug: Lamivudine
- Telbivudine (Experimental): Telbivudine treatment from 28 weeks of pregancy to week 4 of postpartum for mothers and standrd immunoprophylaxis to their infants
  Interventions: Drug: Telbivudine

INTERVENTIONS:
Drug: Telbivudine — About 300 mothers with no treatment observedfrom 28 weeks of pregnancy to the week 4 of postpartun
  Arms: Telbivudine
Drug: Lamivudine — About 300 mothers treated with lamivudine or telbivudine from 28 weeks of pregancy to the week 4 of postpartum
  Arms: Lamivudine

SUMMARY:
To explore the antiviral effect of nucleoside analogue in late pregnancy and the safety of the antiviral drug to fetus.To establish the best therapy strategy to pregnant women with high level of HBV DNA.

DETAILED DESCRIPTION:
Telbivudine and Lamivudine,a preganancy category B medication,reduces HBV DNA and normalizes serum ALT in chronic hepatitis B patients with few adverse effects.Two aspects on the drug use in pregnancy will be evaluated prospectively in this study.

ELIGIBILITY:
Inclusion Criteria:

HBeAg+CHB pregnant woman gestational age 28 weeks HBV-DNA>log10 copies/ml

Exclusion Criteria:

co-infection with hepatitis A,C,D,E or HIV evidence of hepatocellular carcinoma decompensated liver disease or significant co-morbidity concurrent treatment with immune-modulators,cytotoxic drugs,or steroids clinical signs of threatened miscarriage in early prenancy evidence of fetal deformity by ultrasound examination the biological father of the child had CHB

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 700 (Actual)
Dates: Start 2009-03; Primary Completion 2012-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The data on its tolerability and safety in HBeAg+ pregnant woman with HBV DNA>6log10 copies/Ml during late pregnancy and infants | perinatal to 28 weeks after infant delivery
Its efficacy in the reduction of HBV vertical transmission rate | perinatal to 28 weeks after infant delivery

SECONDARY OUTCOMES:
Maternal DNA reduction,ALT normalization, and loss/seroconversion of HBeAg or HBsAg | perinatal to 28 weeks of postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Hua Zhang, MD, Principal Investigator — Beijing YouAn Hospital